CLINICAL TRIAL: NCT03489889
Title: Development of Ursodeoxycholic Acid 300 mg at Hospital Das Clinicas of the University of São Paulo School of Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Cleuber Esteves Chaves, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Gastro FMUSP
Record Dates: First submitted 2018-01-12; First posted 2018-04-06 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Ursodeoxycholic Acid; Primary Biliary Cirrhosis
Keywords: Liver Cirrhosis, Biliary; Ursodeoxycholic Acid
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- capsule (Experimental): pharmaceutical form: capsule ursodeoxycholic acid 300 mg 13-15mg/kg day 3 months
  Interventions: Drug: Ursodeoxycholic Acid 300mg capsule
- tablet (Experimental): pharmaceutical form: tablet ursodeoxycholic acid 300 mg 13-15mg/kg day 3 months
  Interventions: Drug: Ursodeoxycholic Acid 300mg tablet

INTERVENTIONS:
Drug: Ursodeoxycholic Acid 300mg tablet — Cross-over study: Ursodeoxycholic Acid 300mg tablet and after Ursodeoxycholic Acid 300mg capsule
  Arms: tablet
Drug: Ursodeoxycholic Acid 300mg capsule — Cross-over study: Ursodeoxycholic Acid 300mg capsule and after Ursodeoxycholic Acid 300mg tablet
  Arms: capsule

SUMMARY:
A manipulation and an integral part of the pharmaceutical practice, where, in addition to the supply of medicines and personalized products, they represent an alternative to the therapeutic schemes, manipulating drugs of almost all of them as therapeutic categories.

One of the products and ursodeoxycholic acid, commercially known as Ursacol, a bile acid physiologically present in human bile, approved by Agência Nacional de Vigilância Sanitária (ANVISA), among several indications, for the treatment of the symptomatic form of primary biliary cholangitis, autoimmune etiology and predominant incidence in female.

This is a prospective, cross-over, interventional and open-label study, where patients attending the inclusion and exclusion criteria are attended by the Instituto Central do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (ICHC-FMUSP) Pharmacy Division in the Pharmaceutical Care sector.

As patient information as well as the prescribed drugs, compiled by a data collection instrument from the ICHC-FMUSP Pharmacy Division and a semi-structured questionnaire.

DETAILED DESCRIPTION:
The therapeutic efficacy of Ursodeoxycholic Acid 300 mg tablet and capsules was measured comparing the liver enzyme parameters: alkaline phosphatase, gamma glutamyl transferase, alanine aminotransferase, aspartate aminotransferase and total bilirubin in three times: before treatment begins, in the middle of treatment and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Primary biliary cholangitis (PBC) was diagnosed when at least two of the following three criteria: histologically proven early stage PBC; positive Anti-mitochondrial antibody (AMA) (titer >1:40) and alkaline phosphatase >1.5 times upper limit of normal at any time since diagnosis.
* Patients had to be on ursodeoxycholic acid for at least 6 months.
* Patients should be able to understand and ready to sign the informed consent form.

Exclusion Criteria:

* Patients not adherent to treatment with reference medicine.
* Known intolerance to the study drugs.
* Patients who withdrew their agreement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy between capsule and tablet | up to 12 months
  Compare the liver enzyme parameters (alkaline phosphatase, alanine aminotranferase, aspartate aminotransferase, gamma glutamyl transferase and total bilirubin) in three different moments:before the treatment, between the treatment and at the end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Nakano LA, Cancado ELR, Chaves CE, Madeira MCV, Katayose JT, Nabeshima MA, Fossaluza V, Uhrigshardt GG, Liting Z, Pinto VB, Carrilho FJ, Ono SK. A randomized crossover trial to assess therapeutic efficacy and cost reduction of acid ursodeoxycholic manufactured by the university hospital for the treatment of primary biliary cholangitis. BMC Gastroenterol. 2020 Aug 5;20(1):253. doi: 10.1186/s12876-020-01399-5. PMID 32758152